CLINICAL TRIAL: NCT01521468
Title: Prospective Comparison of Cardiac PET/CT, SPECT/CT Perfusion Imaging and CT Coronary Angiography With Invasive Coronary Angiography
Brief Title: Comparison of Cardiac Imaging Techniques for Diagnosing Coronary Artery Disease
Acronym: PACIFIC
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Paul Knaapen, MD, PhD, Amsterdam UMC, location VUmc
Other Study IDs: NL33941.029.10; 2011/209 (Other: Medical Ethical Committee VU University Medical Center)
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Diagnostic accuracy; CT coronary angiography; Positron emission tomography; Single photon emission tomography; Noninvasive techniques; Cardiac catheterization; Fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and whole blood.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A large number of cardiac catheterizations are performed each year, primarily to diagnose heart disease. However, a cardiac catheterization is an invasive procedure which is associated with serious complications such as heart infarction, stroke, and death. Therefore, there is a need for non-invasive procedures to diagnose coronary heart disease. The purpose of this study is, therefore, to assess the diagnostic accuracy of non-invasive cardiac imaging modalities for the detection of heart disease in patients presenting for the first time to the cardiologist with chest pain.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains the leading cause of morbidity and mortality in Western civilized countries. Early detection of CAD allows optimal therapeutic management in order to decrease morbidity and mortality. In the Netherlands 80,000 invasive coronary angiographies are performed each year. Invasive coronary angiography (ICA), particularly in conjunction with fractional flow reserve (FFR) measurements, is considered the gold standard in diagnosing and evaluating the severity of CAD in the current era. FFR measurements during ICA are useful in determining whether a coronary stenosis is functionally important. An FFR < 0.80 is considered abnormal, reflecting a hemodynamic significant coronary stenosis. ICA has superior spatial and temporal resolution compared with non-invasive imaging techniques. However, ICA is an invasive procedure which is associated with a low, though significant, complication rate including bleeding, coronary artery dissections, cerebral embolism, cardiac arrhythmias, myocardial infarction and death. Moreover, ICA provides only limited information on the presence of atherosclerotic plaques not associated with luminal stenosis. Furthermore, conventional catheter angiography without the advent of FFR measurements, is not able to provide information about the hemodynamic significance of a significant luminal stenosis (≥ 70%), i.e. whether a coronary artery stenosis is leading to myocardial perfusion abnormalities. Therefore, there is a need for non-invasive imaging techniques for diagnosing and evaluating the hemodynamic significance of CAD. Non-invasive techniques can serve as a gatekeeper for invasive coronary angiographies in order to decrease the number of purely diagnostic invasive angiographies and associated morbidity and mortality. The detection and management of cardiovascular disease increasingly utilize non-invasive cardiac imaging in patients with suspected or known CAD. By more accurately identifying patients who are eligible for coronary revascularization with the use of non-invasive cardiac imaging, the number of unnecessary invasive diagnostic coronary angiographies can be decreased.

Study design

Positron emission tomography:

PET images will be acquired using a Gemini Time-of-Flight (TF) 64 scanner (Philips Healthcare, Best, The Netherlands). Quantitative myocardial perfusion at rest and during hyperemia in ml -1. min -1. g -1 of myocardial tissue will be measured using oxygen-15-labelled water (H215O). Pharmacological stress is induced by infusion of adenosine intravenously at a rate of 140 µg/kg/min. Two minutes after the start of adenosine vasodilation reaches a steady state and H215O will be given intravenously as a bolus followed with the start of a 6-minutes emission scan. Directly after the PET sequence, a low dose CT attenuation scan (CTAC) is acquired after which the infusion of adenosine is terminated. Technetium-99m sestamibi is injected intravenously after the second CTAC scan. A stress SPECT-scan is performed 45 minutes after the stress PET scan.

Single photon emission computed tomography:

SPECT imaging will be performed according to standard clinical protocols for myocardial perfusion imaging. All patients will undergo SPECT-imaging(Symbia T2, Siemens, The Hague, The Netherlands) on a during hyperaemia induced by infusion of adenosine at a rate of 140mcg/kg/min, using a dose of 400 megabecquerel (MBq) of Technetium (99mTc) tetrofosmin. Tetrofosmin will be administered during adenosine induced stress during the time of the PET stress perfusion scan. Directly after the stress SPECT-sequence, a low dose CT-attenuation scan (CTAC) will be performed. A SPECT- rest imaging scan will be performed 72 hours after the stress SPECT scan on the day of the catheterization.

Computed tomography:

Patients will undergo a coronary calcium score (CTCAC) and CT coronary angiography scan on a 256-slice CT scanner (Philips Brilliance iCT, Philips Healthcare, Best, the Netherlands). Prospective ECG-gating (Step & Shoot Cardiac, Philips Healthcare, Best, The Netherlands) at 75 % of the R-R interval will be performed in order to minimize radiation burden.

Invasive coronary angiography:

ICA will be performed via a transfemoral of transradial approach according to the standard procedure. Iodized contrast will be given intracoronary during the procedure to evaluate the coronary artery lumen. The operator and an interventional cardiologist blinded to the findings obtained with non-invasive imaging will evaluate the ICA images. ICA imaging will be performed with a biplane or monoplane cardiovascular X-ray system (Allura Xper FD 10/10, Philips Healthcare, Best, The Netherlands) in at least two orthogonal directions. After primary coronary angiography, FFR will be measured in all coronary arteries, using a 0.014-inch sensor tipped guide wire. A stenosis with a FFR < 0.80 will be considered as a hemodynamic significant stenosis. Clinical decision making will be based on the findings obtained with ICA and FFR measurements and will be made by the interventional cardiologist.

ELIGIBILITY:
Inclusion Criteria:

* First presentation to cardiologist with suspected coronary artery disease
* No documented prior history of coronary artery disease
* Intermediate pre-test likelihood for coronary artery disease as defined by Diamond and Forrester criteria
* Clinically referred for invasive coronary angiography
* Age above 40 years

Exclusion Criteria:

* History of severe chronic obstructive pulmonary disease (COPD) or chronic asthma
* Pregnancy
* Renal failure ( i.e. estimated glomerular filtration rate < 45 mL/min)
* Use of sildenafil (Viagra) or dipyridamole (Persantin) that can not be terminated.
* Contra-indications for β-blockers
* Allergic reaction to iodized contrast
* Concurrent or prior (within last 30 days) participation in other research studies using investigational drugs
* Claustrophobia
* Significant co-morbidities
* Atrial fibrillation, second or third degree atrioventricular block
* Tachycardia
* Acute myocardial infarction
* Heart failure
* Left ventricle ejection fraction estimated < 50%
* Cardiomyopathies
* Previous radiation exposure in the diagnostic work-up
* Subjects intended for short-term medical treatment or an invasive coronary intervention
* No informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic of the VU University Medical Center hospital in Amsterdam.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Head to head comparison between hybrid SPECT/CTCA and PET/CTCA | Invasive coronary angiography + fractional flow reserve measurements within 1 week of the initial scans
  A head-to-head comparison will be performed to assess the diagnostic accuracy of stress hybrid PET/CTCA and hybrid SPECT/CTCA for the detection of obstructive coronary artery disease as defined by invasive coronary angiography in combination with fractional flow reserve measurements.
Non-invasive imaging for risk stratification | Ten years
  To determine the prognostic value of CTCA, SPECT, quantitative PET, hybrid SPECT/CTCA and PET/CTCA for predicting cardiac death and nonfatal myocardial infarction.
Improving prognostication | Ten years
  To compare the ability and incremental value of non-invasive stand-alone and cardiac hybrid imaging over clinical, historical and exercise test data for the prediction of all cause mortality.
Diagnostic accuracy of CTCA, SPECT and PET | Invasive coronary angiography + fractional flow reserve measurements within 1 week of the initial scans
  Determining the diagnostic accuracy of stand-alone cardiac imaging modalities

SECONDARY OUTCOMES:
Risk stratification | Ten years
  To determine the incremental prognostic value of several biomarkers over non-invasive imaging, clinical, historical and exercise test data to predict overall mortality, nonfatal myocardial infarction, revascularization and hospitalization for chest pain or heart failure.
Risk stratification | > 6 months
  To compare the predictive and incremental value of stand-alone and cardiac hybrid imaging imaging over clinical, historical and exercise test data for the prediction of a composite endpoint including cardiac death, nonfatal myocardial infarction, late referral to revascularization, or late hospitalization for chest pain or heart failure.
Risk stratification | > 6 months
  To compare the predictive and incremental value of several biomarkers over non-invasive imaging, clinical, historical and exercise test data for the prediction of a composite endpoint including cardiac death, nonfatal myocardial infarction, late referral to revascularization, or late hospitalization for chest pain or heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Knaapen, MD, PhD, Principal Investigator — VU University Medical Center, ICaR-VU
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Background] Kajander S, Joutsiniemi E, Saraste M, Pietila M, Ukkonen H, Saraste A, Sipila HT, Teras M, Maki M, Airaksinen J, Hartiala J, Knuuti J. Cardiac positron emission tomography/computed tomography imaging accurately detects anatomically and functionally significant coronary artery disease. Circulation. 2010 Aug 10;122(6):603-13. doi: 10.1161/CIRCULATIONAHA.109.915009. Epub 2010 Jul 26. PMID 20660808
- [Background] Di Carli MF, Hachamovitch R. New technology for noninvasive evaluation of coronary artery disease. Circulation. 2007 Mar 20;115(11):1464-80. doi: 10.1161/CIRCULATIONAHA.106.629808. No abstract available. PMID 17372188
- [Background] Gaemperli O, Husmann L, Schepis T, Koepfli P, Valenta I, Jenni W, Alkadhi H, Luscher TF, Kaufmann PA. Coronary CT angiography and myocardial perfusion imaging to detect flow-limiting stenoses: a potential gatekeeper for coronary revascularization? Eur Heart J. 2009 Dec;30(23):2921-9. doi: 10.1093/eurheartj/ehp304. Epub 2009 Aug 14. PMID 19684023
- [Background] Schuijf JD, Wijns W, Jukema JW, Atsma DE, de Roos A, Lamb HJ, Stokkel MP, Dibbets-Schneider P, Decramer I, De Bondt P, van der Wall EE, Vanhoenacker PK, Bax JJ. Relationship between noninvasive coronary angiography with multi-slice computed tomography and myocardial perfusion imaging. J Am Coll Cardiol. 2006 Dec 19;48(12):2508-14. doi: 10.1016/j.jacc.2006.05.080. Epub 2006 Nov 28. PMID 17174190
- [Background] Knaapen P, de Haan S, Hoekstra OS, Halbmeijer R, Appelman YE, Groothuis JG, Comans EF, Meijerink MR, Lammertsma AA, Lubberink M, Gotte MJ, van Rossum AC. Cardiac PET-CT: advanced hybrid imaging for the detection of coronary artery disease. Neth Heart J. 2010 Feb;18(2):90-8. doi: 10.1007/BF03091744. PMID 20200615
- [Background] Pijls NH, De Bruyne B, Peels K, Van Der Voort PH, Bonnier HJ, Bartunek J Koolen JJ, Koolen JJ. Measurement of fractional flow reserve to assess the functional severity of coronary-artery stenoses. N Engl J Med. 1996 Jun 27;334(26):1703-8. doi: 10.1056/NEJM199606273342604. PMID 8637515
- [Background] Levin DC. Invasive evaluation (coronary arteriography) of the coronary artery disease patient: clinical, economic and social issues. Circulation. 1982 Nov;66(5 Pt 2):III71-9. PMID 7127709
- [Background] Pazhenkottil AP, Nkoulou RN, Ghadri JR, Herzog BA, Kuest SM, Husmann L, Wolfrum M, Goetti R, Buechel RR, Gaemperli O, Luscher TF, Kaufmann PA. Impact of cardiac hybrid single-photon emission computed tomography/computed tomography imaging on choice of treatment strategy in coronary artery disease. Eur Heart J. 2011 Nov;32(22):2824-9. doi: 10.1093/eurheartj/ehr232. Epub 2011 Jul 30. PMID 21804107
- [Background] Gaemperli O, Bengel FM, Kaufmann PA. Cardiac hybrid imaging. Eur Heart J. 2011 Sep;32(17):2100-8. doi: 10.1093/eurheartj/ehr057. Epub 2011 Mar 15. PMID 21406437
- [Background] Pazhenkottil AP, Nkoulou RN, Ghadri JR, Herzog BA, Buechel RR, Kuest SM, Wolfrum M, Fiechter M, Husmann L, Gaemperli O, Kaufmann PA. Prognostic value of cardiac hybrid imaging integrating single-photon emission computed tomography with coronary computed tomography angiography. Eur Heart J. 2011 Jun;32(12):1465-71. doi: 10.1093/eurheartj/ehr047. Epub 2011 Feb 14. PMID 21320906
- [Derived] Wilgenhof A, Jukema RA, Driessen RS, Danad I, Raijmakers PG, van Royen N, van Nunen LX, Collet C, de Waard GA, Knaapen P. The effect of hydrostatic pressure on invasive coronary pressure measurements: Comparison with [15O]H2O-positron emission tomography flow data. Catheter Cardiovasc Interv. 2024 Nov;104(5):980-989. doi: 10.1002/ccd.31215. Epub 2024 Sep 11. PMID 39258435
- [Derived] Arai AE. Why Should We Quantify Stress Myocardial Perfusion CMR? JACC Cardiovasc Imaging. 2024 Mar;17(3):266-268. doi: 10.1016/j.jcmg.2023.08.015. Epub 2023 Oct 18. No abstract available. PMID 37855801
- [Derived] Lin A, van Diemen PA, Motwani M, McElhinney P, Otaki Y, Han D, Kwan A, Tzolos E, Klein E, Kuronuma K, Grodecki K, Shou B, Rios R, Manral N, Cadet S, Danad I, Driessen RS, Berman DS, Norgaard BL, Slomka PJ, Knaapen P, Dey D. Machine Learning From Quantitative Coronary Computed Tomography Angiography Predicts Fractional Flow Reserve-Defined Ischemia and Impaired Myocardial Blood Flow. Circ Cardiovasc Imaging. 2022 Oct;15(10):e014369. doi: 10.1161/CIRCIMAGING.122.014369. Epub 2022 Oct 13. PMID 36252116
- [Derived] de Waard GA, Danad I, Petraco R, Driessen RS, Raijmakers PG, Teunissen PF, van de Ven PM, van Leeuwen MAH, Nap A, Harms HJ, Lammertsma AA, Davies JE, Knaapen P, van Royen N. Fractional flow reserve, instantaneous wave-free ratio, and resting Pd/Pa compared with [15O]H2O positron emission tomography myocardial perfusion imaging: a PACIFIC trial sub-study. Eur Heart J. 2018 Dec 7;39(46):4072-4081. doi: 10.1093/eurheartj/ehy632. PMID 30452609